CLINICAL TRIAL: NCT01779011
Title: Suivi et Traitement du Traumatisme Des Membres en Cas d'Afflux Massif de blessés Dans Les Contextes Difficiles
Brief Title: Monitoring and Treatment of Extremity Trauma for Mass Casualties in Difficult Contexts
Acronym: SuTra²
Status: Completed | Type: Observational
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Lille Economie Management UMR CNRS 8157 (Unknown); National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: SuTra² (Suivi et Traitement du
Record Dates: First submitted 2012-12-15; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Wounds and Injuries; Traumatic Amputation
MeSH Terms: conditions — Wounds and Injuries; Amputation, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A cohort post amputation: Those patients undergoing either traumatic amputation or surgical amputation of limb
- A cohort post limb conserving surgery: Patients whose surgical management involved conservation of their injured limb

SUMMARY:
The prospective cohort study, SuTra2, assesses the functional and socio-economic status of patients who were operated on for a severe limb injury resulting in amputation or limb preservation 1 and 2 years after the 2010 Haiti earthquake.

ELIGIBILITY:
Inclusion Criteria:

* Patients, with limb injuries due to the earthquake,
* Who underwent limb surgery, which ended up in limb amputation or limb conservation.

Exclusion criteria :

* Limb injury not related to the earthquake
* No surgery for the limb injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited by phone from databases issued by:
  * A surgical clinic, The Clinique Lambert (Pétion-Ville, Haiti),
  * Two non-governmental organizations
    * Handicap International (HI)
    * Bangladesh Rural Advancement Committee (BRAC),
  * A local organization l'Union des Jeunes Victimes du Séisme (UJVS)
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction with Musculoskeletal functional recovery | 2 years

SECONDARY OUTCOMES:
Employment status | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine Delauche, MD, Principal Investigator — Alliance for International Medical Action
Locations (1):
- ALIMA, Port-au-Prince, Port-au-Prince, Haiti

REFERENCES:
- See also: ALIMA website with links within to full study protocol in French — http://www.alimaong.org